CLINICAL TRIAL: NCT00797550
Title: Use of TRC Autologous Bone Marrow Cells in Posterolateral Lumbar Spine Fusion
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated early for business reasons (not safety reasons).
Sponsor: Vericel Corporation (Industry)
Responsible Party: Elmar Burchardt, MD, PhD, Aastrom Biosciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-55-0509-1
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Single Level Posterolateral Spinal Fusion
Keywords: posterolateral spine fusion; bone graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): The Control arm of the study will receive bone autograft.
  Interventions: Procedure: Autologous bone graft
- Treatment (Experimental): The Treatment arm of the study will receive single level posterolateral spinal fusion between L1 to S1 levels with implantation of BRC product.
  Interventions: Biological: Bone Repair Cells (BRCs)

INTERVENTIONS:
Biological: Bone Repair Cells (BRCs) — BRCs will be administered during spine fusion surgery
  Other Names: autologous bone marrow cells
  Arms: Treatment
Procedure: Autologous bone graft
  Arms: Control

SUMMARY:
The hypothesis is that Aastrom TRC autologous bone marrow tissue "grafts" can be safely used to promote bone healing as part of a single level posterolateral spine fusion surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-75 years of age
* Identified as eligible for elective surgery for single (1) level, posterolateral spinal fusion between L1 and S1 in which the spine stabilization is accomplished by pedicle screws and rod.
* Male patients and female patients (not pregnant or lactating). Patients should use an appropriate form of contraception while participating in the study.
* Patients able to give informed consent.
* Normal organ and marrow function

Exclusion Criteria:

* Patients with hypophosphatasia, primary or secondary hyperparathyroidism caused by chronic renal insufficiency or osteomalacia.
* Patients with osteoporotic vertebral fractures.
* Patients with a prior spinal fusion at the level to be treated.
* Concomitant use of BMP, or devices containing BMP, or electronic growth stimulators.
* Any active infection of any clinical significance will be excluded from the study.
* Positive for HIV, HTLV and/or syphilis.
* Active Hepatitis B, or Hepatitis C infection at the time of enrollment.
* Known allergies to protein products (horse or bovine serum, or porcine trypsin) used in the ex-vivo cell production process.
* Patients who require systemic corticosteroid therapy after surgery.
* Pregnancy or lactation; positive of hCG.
* Body Mass Index (BMI) of 40 Kg/m2 or greater.
* Patients unable to tolerate general anesthesia defined as an ASA criteria of >2.
* Patients with poorly controlled diabetes mellitus (HbA1C >7%).
* Rationale for Exclusion of Certain Study Candidates

  1. Patients with other diseases are excluded to avoid confounding factors that might impact evaluation of safety and efficacy of TRC cell therapy in posterolateral spine fusion.
  2. More extensive surgery requiring more than one (1) level fusion is contraindicated in this study, to avoid confounding factors that might impact evaluation of safety and efficacy of TRC cell therapy.
* In the opinion of the investigator, the patient is unsuitable to cellular therapy or unable to continue with this study.
* Patients that drink more than 2 alcoholic drinks per day or have a history of illicit drug use at the time of enrollment shall not be enrolled in the study.
* Patient known to be non-euthyroid at baseline.
* Patients undergoing active cancer therapy.
* Bisphosphonate Therapy

  1. Patients that have undergone bisphosphonate therapy within the last 10 years.
  2. Initiation of bisphosphonate therapy in patients during this study is prohibited.
* Patients with a known diagnosis of osteoporosis with recorded BMD less than -2.5.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to confirm that the TRC product, when used as a bone graft, is safe for use in posterolateral lumbar spinal fusion surgery, on the basis of defined radiographic evidence of bone fusion. | Throughout duration of study

SECONDARY OUTCOMES:
To assess the relative efficacy of TRC graft compared to autologous vertebral bone graft based on the frequency and extent of callus or bone bridging between the adjacent decorticated vertebral processes on each side of the vertebrae. | Imaged by CT at 6 months after surgery
To assess surgeon's evaluation of radiographic healing at the site of surgery based on flexion and extension radiographs, as well as 2AP and lateral radiographs, and of clinical resolution | Baseline, Month 6 and Month 12
To assess reduction in pain scores at site of back surgery | First 3 months post-treatment
To assess use of prescription and non-prescription pain control and other drugs in treatment patients as compared to control patients | Throughout duration of study
To assess restoration of function for return to activities of normal daily living | Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Harry Herkowitz, MD, Principal Investigator — Corewell Health East